CLINICAL TRIAL: NCT06899841
Title: Effect of Different Doses of Dexmedetomidine Added to Local Anesthetic in Sonographic Guided Erector Spinae Plane Block for Pain Management After Renal Surgeries : Randomized Clinical Trial
Brief Title: Dexmedetomidine in Sonographic Guided Erector Spinae Plane Block
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Faisal, dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-2024-200943
Record Dates: First submitted 2025-03-16; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose dex (Experimental): 0.5 mic/kg of dexmedetomidine administered
  Interventions: Drug: Dexmedetomidine
- intermediate dose dex (Experimental): 0.75 mic/kg of dexmedetomidine administered
  Interventions: Drug: Dexmedetomidine
- high dose dex (Experimental): 1 mic/kg of dexmedetomidine administered
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — different doses of dexmedetomidine added to bupivacaine in erector spinae plane block

SUMMARY:
to investigate the postoperative analgesic effect of dexmedetomidine addition with different doses as an adjuvant to bupivacaine to Erector spinae plane block after renal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years.
* Both sexes, males and females.
* Patients with the American Society of Anesthesiologists (ASA) physical status I/II.
* Body mass index (BMI) of 18-35 kg/m2
* Patients scheduled for elective Renal or Percutaneous Nephrolithotomy.

Exclusion Criteria:

* Patients under 18 years.
* Patient refusal of nerve block.
* Infection at the site of injection.
* Coagulopathy.
* Allergy to used medications.
* Psychiatric disorder or chronic pain syndromes.
* Chronic opioid use or substance abuse.
* Quadriplegic patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
postoperative analgesic duration | 24 hours
  postoperative analgesic duration with each dose

SECONDARY OUTCOMES:
Pain score | 24 hours
  severity of pain using visual analogue pain score
side effects | 24 hours
  as hemodynamic effect as (hypotension, bradycardia), nausea and vomiting.
dynamic pain score | 24 hours
  Dynamic visual analogue pain score (pain with cough, deep breath, and movement)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No